CLINICAL TRIAL: NCT06618781
Title: Perioperative Effects of Lateral Quadratus Lumborum Block in Percutaneous Transhepatic Cholangiography: Prospective Observational Study
Brief Title: Perioperative Effects of Lateral Quadratus Lumborum Block in Percutaneous Transhepatic Cholangiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Seyyid Furkan Kına, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEŞH-EK1-2024-0061
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2024-10

CONDITIONS: Opioid Consumption; Visual Analog Score; Demographic Data; Rescue Analgesic Status and Time
Keywords: Percutaneous transhepatic cholangiography; Quadratus lumborum block; Interventional Radiology

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group sedation (Active Comparator): Preoperatively, 2 mg intravenous midazolam was administered to the patients. Intravenous 0.5 mg/kg propofol and 0.5 mcg/kg fentanyl were used for induction. Intravenous 0.5-1 mg/kg propofol was administered to provide an intraoperative bispectral index of 40-60, and when the Vizel analog score was >4, intravenous 0.1-1 mcg/kg remifentanil was administered. Postoperatively, 1 g paracetamol was routinely administered. When the Vizel analog score was >4, 50 mg dexketoprofen was administered as a rescue analgesic. Postoperative 2nd, 6th, 12th and 24th hour visual analog scores of the patients were recorded.
  Interventions: Procedure: Sedation
- Group sedation+ Quadratus Lumborum Block (Active Comparator): Before the procedure, the patient was placed in the left lateral position and a Quadratus Lumborum Block was applied at the thoracic 8-10 level. A total of 20 cc blocking fluid consisting of 14 cc of 0.5% bupivacaine and 6 cc of 2% lidocaine was used for the block. A minimum of 30 minutes was waited after the block. 2 mg of intravenous midazolam was administered before being taken to the operating room. Intravenous 0.5 mg/kg propofol and 0.5 mcg/kg fentanyl were used for induction. Intravenous 0.5-1 mg/kg propofol was administered to provide an intraoperative bispectral index of 40-60, and intravenous 0.1-1 mcg/kg remifentanil was administered when the Vizel analog score was > 4. Postoperatively, 1 g of paracetamol was routinely administered. When the Vizel analog score was > 4, 50 mg of dexketoprofen was administered as a rescue analgesic. Postoperative 2nd, 6th, 12th and 24th hour visual analog scores of the patients were recorded.
  Interventions: Procedure: Sedation + Quadratus Lumborum Block

INTERVENTIONS:
Procedure: Sedation — Preoperatively, 2 mg intravenous midazolam was administered to the patients. Intravenous 0.5 mg/kg propofol and 0.5 mcg/kg fentanyl were used for induction. Intravenous 0.5-1 mg/kg propofol was administered to provide an intraoperative bispectral index of 40-60, and when the Vizel analog score was >4, intravenous 0.1-1 mcg/kg remifentanil was administered.
  Arms: group sedation
Procedure: Sedation + Quadratus Lumborum Block — Before the procedure, the patient was placed in the left lateral position and a Quadratus Lumborum Block was applied at the thoracic 8-10 level. A total of 20 cc blocking fluid consisting of 14 cc of 0.5% bupivacaine and 6 cc of 2% lidocaine was used for the block. A minimum of 30 minutes was waited after the block. 2 mg of intravenous midazolam was administered before being taken to the operating room. Intravenous 0.5 mg/kg propofol and 0.5 mcg/kg fentanyl were used for induction. Intravenous 0.5-1 mg/kg propofol was administered to provide an intraoperative bispectral index of 40-60, and intravenous 0.1-1 mcg/kg remifentanil was administered when the Vizel analog score was >4.
  Arms: Group sedation+ Quadratus Lumborum Block

SUMMARY:
The frequency of non-operating room anesthesia (ADA) applications is increasing and has gained an important place in anesthesia practice. Percutaneous transhepatic cholangiography (PTC) procedures applied in interventional radiology are also examples of ADA. It is frequently applied for both diagnostic and therapeutic purposes in cases where obstruction is observed in the bile ducts for any reason. Providing a balanced and comfortable anesthesia during PTC procedures reduces postoperative complications and increases patient and clinician satisfaction. General anesthesia, sedoanesthesia and regional anesthesia can be applied in PTCs. Due to the perioperative complications and undesirable side effects of general anesthesia, it is not the first choice in PTCs. Sedoanesthesia and regional anesthesia are widely applied in PTCs. Postoperative pain is the most important parameter affecting patient satisfaction in this surgery. Inadequate treatment of postoperative pain can reduce the quality of life and cause chronic pain syndromes. In order to effectively combat pain; regional methods are frequently used in addition to intravenous analgesics. For PTC patients, Erector Spinae Plane Block, Quadratus Lumborum Block (QLB) and Subcostal TAP block can be applied covering the T6-L1 dermatome. Since the pain in PTC patients is of visceral and somatic origin, the one with the highest analgesic efficacy is QLB. 4 different techniques of QLB have been defined in the literature and these techniques are; lateral, posterior, anterior transmuscular and intramuscular. Local anesthetic spread is relatively low in the intramuscular technique, while the risk of complications is high in the transmuscular technique. However, lateral and posterior techniques are not superior to each other, and the experience of the clinician is effective in the selection of the technique. The mechanism of action of QLB depends on ipsilateral paravertebral and epidural local anesthetic spread. There are studies in the literature that QLB is used in trunk and abdominal surgeries; provides effective analgesia and reduces the amount of opioid consumed. Due to all these effects, interest in QLB is increasing and its use is becoming widespread. Lateral QLB application: In the left lateral decubitus position, the curvelinear (5-1 MHz) USG probe is placed in the iliac crest and subcostal area at the level of T8-10. Then, the probe is directed posteriorly and cranially to provide detailed visualization of the anterolateral surface of the vertebral body with the transverse process. The probe is slightly tilted to identify the psoas major, quadratus lumborum and erector spinae muscles. The typical image of these 3 muscles forms a three-leaf 'clover' pattern. With the lateral approach, at the point where the transverse abdominis muscle ends, hydrodissection is performed with 2 cc physiological serum to the lateral side of the quadratus lumborum to confirm the location. Then, a total of 20 cc blocking fluid consisting of 14 cc of 0.5% bupivacaine and 6 cc of 2% lidocaine is injected into this area. The blocking fluid is applied in divided doses of 5 cc with intermittent negative aspiration. In our clinic, multimodal anesthesia/analgesia method is preferred in patients undergoing PTC procedure. Peripheral nerve blocks (for all patients who are suitable and accept) are routinely used together with intravenous analgesic agents. The applied block aims to reduce the amount of opioid consumed perioperatively, faster postoperative recovery, lower postoperative VAS scores, lower postoperative analgesia consumption and earlier mobilization. QLB is routinely applied in suitable patients undergoing PTC. Patients who are subjected to sedoanesthesia and those who are subjected to QLB together with sedoanesthesia will be included in the study. The anesthesiologist who provides the anesthesia management of the patients and the anesthesiologist who monitors the patient's pain will be different individuals.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18-80
* Those with ASA score I-II-III
* Those with body mass index (BMI) between 18-40
* Patients who underwent sedoanesthesia and sedoanesthesia and QLB for PTC procedure

Exclusion Criteria:

* Those under 18 and over 80
* Those with ASA score IV and above
* Those with advanced co-morbidities
* Those with a history of bleeding diathesis
* Patients with an infection in the area where the block will be performed
* Those with a BMI below 18 and above 40
* Patients who underwent surgery under emergency conditions
* Those who are pregnant
* Those with opioid and local anesthetic allergies-
* Those with chronic pain syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-10-11 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Intraoperative remifentanil consumption. | Intraoperative period
  Intraoperative remifentanil consumption will be recorded.

SECONDARY OUTCOMES:
Intraoperative propofol consumption. | Intraoperative period
  Intraoperative propofol consumption will be recorded.
Pain Scores | 24 hours after surgery
  Pain will be assessed at rest and coughing using the visual analog scale on a scale form 0 (no pain) to 10 (worst pain). Pain assessment will be done at the 2nd, 6th, 12th, 24th hours after the surgery. Visual analog scale 10 (worst) severe, unbearable pain; 0 (best) no pain.
Postoperative rescue analgesic | During the postoperative 24 hours
  atients with a VAS score of 4 and above will receive rescue analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Seyyid Furkan Kına, MD, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Altındağ, Ankara, Turkey (Türkiye)